CLINICAL TRIAL: NCT03614169
Title: Direct HIS-pacing as an Alternative to Biventricular Pacing in Symptomatic Heart Failure Patients With Severely Reduced LVEF and a True Left Bundle Branch Block
Brief Title: Direct HIS-pacing as an Alternative to BiV-pacing in Symptomatic HFrEF Patients With True LBBB
Acronym: HISalternative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Vinther, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIS-alternative
Record Dates: First submitted 2018-07-29; First posted 2018-08-03 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Left Bundle-Branch Block
Keywords: HIS-pacing; Biventricular pacing
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct HIS-pacing (Experimental): In this arm a right ventricular (RV) lead or implantable cardioverter defibrillator (ICD) lead is placed first and then implantation of a HIS-pacing lead is attempted. If it is not possible to find and pace HIS or it is not possible to correct the LBBB, a left ventricular (LV) lead is implanted instead.
  Interventions: Procedure: Implantation of a HIS-pacing lead
- Biventricular pacing (Active Comparator): In this arm an RV-lead or ICD-lead is placed first and then implantation of a LV-pacing lead is attempted. If this is not possible due to anatomical difficulties (no coronary sinus (CS) access, no available branches other than v cordis anterior or v cordis media) or electrical difficulties (no capture below 4 V at 1.0 msec or phrenic nerve stimulation < 2x pacing threshold)
  Interventions: Procedure: Implantation of a LV-pacing lead

INTERVENTIONS:
Procedure: Implantation of a HIS-pacing lead — This intervention is attempted first
  Arms: Direct HIS-pacing
Procedure: Implantation of a LV-pacing lead — This intervention is attempted first
  Arms: Biventricular pacing

SUMMARY:
The present study will randomize 50 symptomatic heart failure patients with severely reduced left ventricular ejection fraction (LVEF) and a true left bundle branch block to either direct HIS-pacing or biventricular pacing and follow them for at least six months. The outcome is how often it is possible to achieve HIS-pacing at implant and during follow-up and if HIS-pacing leads to differences in symptoms or measurable clinical parameters as compared to biventricular pacing.

DETAILED DESCRIPTION:
Biventricular (BiV) pacing is an established treatment of symptomatic heart failure patients with severely reduced left ventricular ejection fraction (HFrEF) and wide QRS due to bundle branch block (BBB) on a 12-lead ECG. BiV pacing is normally achieved with an endocardial pacing lead in the right ventricle and an epicardial lead over the left ventricle situated in a coronary vein. BiV pacing does not correct the BBB but corrects the mechanical dyssynchrony that is a consequence of the BBB. It has been shown to work best on patients with "true" left bundle branch block (LBBB) where the block is due to disease within the conduction system (and not for example left ventricular hypertrophy or scars). Even if the patient is an ideal candidate for BiV pacing it can sometimes be difficult to achieve the best mechanical resynchronization because of anatomic difficulties, high pacing thresholds or phrenic nerve capture.

In recent years it has been demonstrated that the level of block in true LBBB is often within the bundle of HIS and it is possible in many cases to place a pacing lead distally to the site of block and get capture of both right and left bundles thereby "correcting" the BBB and achieve a normal or near-normal QRS complex. If the conduction system is intact distal to the block this mode of pacing leads to complete resynchronization of the ventricles. HIS-pacing can be achieved as either selective HIS-capture where it is only the conduction system that is paced leading to a narrow QRS complex. However, mostly it is achieved with non-selective HIS-capture where both the septal myocardium close to the pacing site and the His-bundle is captured. This leads to a QRS resembling the QRS achieved by selective HIS-capture but preceded by a delta-wave-like deflection which broadens the QRS complex. Since it is only a small part of the septum that is captured early this does not influence the resynchronization of the heart. In some patients HIS-pacing cannot be achieved due to anatomical difficulties that hinders reaching the HIS bundle with the present tools available. In others it is not possible to come distal to the block and recruiting both the left and the right bundle branch.

There is to date no randomized studies between HIS-bundle pacing and BiV pacing in HFrEF patients with LBBB but there are several case reports and retrospective data on successful HIS-bundle pacing in these patients. The present study will randomize 50 patients in a single centre to HIS-pacing or BiV pacing to determine to which extent it is possible to achieve normalization or near-normalization of the QRS with HIS-bundle pacing and what this translates to with regard to symptom relieve, walking distance, echocardiographic measures and N-terminal pro B-type natriuretic peptide (NT-proBNP) levels as compared to BiV pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischaemic or non-ischaemic cardiomyopathy
* LVEF ≤ 35 % as assessed by echocardiography
* New York Heart Association (NYHA) class II-IV despite optimal medical therapy
* Either found eligible for cardiac resynchronization therapy (CRT-P or CRT-D) because of sinus rhythm and "true" LBBB according to Strauss criteria on a 12-lead ECG
* or found eligible for upgrade of an existing pacing system to cardiac resynchronization therapy (CRT-P or CRT-D) because of sinus rhythm and "true" LBBB according to Strauss criteria on a 12-lead ECG or at least 90 % right ventricular pacing in the preceding two months.
* Signed informed consent

Exclusion Criteria:

* Existing biventricular pacing system
* Permanent atrial fibrillation
* Severe kidney failure (eGFR < 30 ml/min)
* Acute myocardial infarction or Coronary By-pass Grafting within the preceding three months
* unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Success rate of obtaining capture of HIS-bundle with narrowing of the QRS-duration | 6 months
  What is the success rate of implanting a pacing lead to the HIS bundle with narrowing of the QRS duration and maintaining this effect during the course of the study

SECONDARY OUTCOMES:
Fall in end-systolic volume > 15% | 6 months
  How many HIS-paced patients as opposed to BiV paced patients have a fall in end-systolic volume > 15 % of the initial value?

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Result] Vinther M, Risum N, Svendsen JH, Mogelvang R, Philbert BT. A Randomized Trial of His Pacing Versus Biventricular Pacing in Symptomatic HF Patients With Left Bundle Branch Block (His-Alternative). JACC Clin Electrophysiol. 2021 Nov;7(11):1422-1432. doi: 10.1016/j.jacep.2021.04.003. Epub 2021 Apr 25. PMID 34167929